CLINICAL TRIAL: NCT04958135
Title: A Phase 1, Randomized, Open-Label, 2-Period, 2-Sequence, 2-Way Crossover Study to Assess the Effect of Food on the Single Dose Pharmacokinetics of Acoramidis in Healthy Participants
Brief Title: Study to Assess the Effect of Food on a Single Dose of Acoramidis in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN2060-HV-101
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Acoramidis; ALXN2060; AG10; Pharmacokinetics; Food Effect; Crossover
MeSH Terms: interventions — attruby

STUDY DESIGN:
Intervention Model Description: This will be a balanced, 2-period, 2-sequence, 2-way crossover study in healthy participants. All participants will receive 1 treatment in each period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Acoramidis (Experimental): Participants will receive acoramidis once each period as a single dose under fasted or fed conditions as follows:
  Period 1: Acoramidis as an immediate-release tablet under fasted conditions.
  Period 2: Acoramidis as an immediate-release tablet under fed conditions.
  There will be a washout period of at least 14 days between acoramidis dosing.
  Interventions: Drug: Acoramidis
- Sequence 2: Acoramidis (Experimental): Participants will receive acoramidis once each period as a single dose under fasted or fed conditions as follows:
  Period 1: Acoramidis as an immediate-release tablet under fed conditions.
  Period 2: Acoramidis as an immediate-release tablet under fasted conditions.
  There will be a washout period of at least 14 days between acoramidis dosing.
  Interventions: Drug: Acoramidis

INTERVENTIONS:
Drug: Acoramidis — Film-coated immediate release oral tablet.
  Other Names: ALXN2060; AG10

SUMMARY:
The purpose of this study is to determine the effect of a high-fat, high-caloric meal on the pharmacokinetics (PK) of acoramidis in healthy adult participants following an oral single dose administration of acoramidis. Blood sampling for PK assessment will include measures for acoramidis and its metabolite, acoramidis acyl glucuronide (acoramidis-AG).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who are healthy as determined by medical evaluation with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory evaluation (hematology, chemistry, urinalysis, and coagulation) that are reasonably likely to interfere with the participant's participation in or ability to complete the study, or to potentially confound interpretation of study results, as assessed by the Investigator.
* Body weight ≥ 50 to ≤ 100 kilograms (kg) and body mass index within the range ≥ 18 to < 32 kg/meter squared for all participants.

Key Exclusion Criteria:

* Evidence of any clinically significant deviation from normal in clinical laboratory evaluations, as determined by the Investigator or designee.
* History of any medical or psychiatric condition or disease that, in the opinion of the Investigator or designee, might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* History or presence of clinically significant hypersensitivity or idiosyncratic reaction to the study interventions or related compounds. History of allergy to other drugs or food will be evaluated by the Investigator or designee on a case by case basis and a decision to enroll will be made by the Investigator or designee.
* Any clinically relevant history or the presence of respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric disease or diseases.
* Disorders of central nervous system, psychiatric disorders, behavioral disturbances (for example, cerebrovascular events, depression, post-traumatic stress disorder, anxiety, bipolar disorder, severe migraine, Parkinson's disease).
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the participant in this study.
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days prior to the first dose of study intervention.
* Female participants who are pregnant, as evidenced by a positive serum pregnancy test result at Screening, or breastfeeding.
* Prior exposure to ALXN2060.
* Major surgery or hospitalization within 90 days prior to dosing on Day 1.
* Use of tobacco in any form (for example, smoking, chewing or vaping), other nicotine-containing products in any form (for example, gum, patch, electronic cigarettes, or vapes), or any recreational inhalational product within 6 months prior to the planned first day of dosing.
* Use of known drugs of abuse within 6 months prior to the planned first day of dosing.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of > 14 units/week for males or > 7 units/week for females. One unit is equivalent to 8 grams of alcohol: a half pint (~240 milliliters [mL]) of beer, one ~4 ounce glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Positive urine drug toxicology screen at Screening or check-in (Day -1).
* Alcohol consumption within 24 hours prior to study intervention administration or positive alcohol breath test at Screening or check-in (Day -1).
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) Of Acoramidis: Fed (Test) Versus Fasted (Reference) Conditions | Up to 336 hours postdose
Area Under The Plasma Concentration Versus Time Curve From Time 0 To The Last Quantifiable Concentration (AUC0-t) For Acoramidis: Fed (Test) Versus Fasted (Reference) Conditions | Up to 336 hours postdose
Area Under The Plasma Concentration Versus Time Curve From Zero To Infinity (AUC0-inf) For Acoramidis: Fed (Test) Versus Fasted (Reference) Conditions | Up to 336 hours postdose

SECONDARY OUTCOMES:
Cmax Of Acoramidis-AG: Fed (Test) Versus Fasted (Reference) Conditions | Up to 336 hours postdose
AUC0-t For Acoramidis-AG: Fed (Test) Versus Fasted (Reference) Conditions | Up to 336 hours postdose
AUC0-inf For Acoramidis-AG: Fed (Test) Versus Fasted (Reference) Conditions | Up to 336 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes